CLINICAL TRIAL: NCT06556264
Title: Determining the Immunologic Impact of Dupilumab on the Unified Airway System in Patients Suffering From Asthma and Chronic Rhinosinusitis With Polyps
Brief Title: Immunologic Impact of Dupilumab in Patients Suffering From Asthma and Chronic Rhinosinusitis With Polyps
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Andrew Thamboo, MD (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor-Investigator, Dr. Andrew Thamboo, MD, Clinical Assistant Professor, St. Paul's Sinus Centre
Organization: St. Paul's Sinus Centre (Other)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H24-00189
Record Dates: First submitted 2024-07-08; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps; Asthma
MeSH Terms: conditions — Asthma | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dupilumab (Active Comparator): 30 subjects undergoing ESS + dupilumab 300 (1-week post-surgery) every 2 weeks + standard of care treatment (INCS + background asthma medication) for 24 weeks
  Interventions: Drug: Dupilumab
- Placebo (Placebo Comparator): 30 subjects undergoing ESS + placebo (1-week post-surgery) every 2 weeks + standard of care treatment (INCS + background asthma medication) for 24 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dupilumab — Dupilumab 300mg every 2 weeks for 24 weeks
  Other Names: dupixent
  Arms: Dupilumab
Other: Placebo — Placebo 300mg every 2 weeks for 24 weeks
  Arms: Placebo

SUMMARY:
The investigators are studying adults who have chronic rhinosinusitis with nasal polyps (CRSwNP) and moderate to severe asthma, and who are undergoing Endoscopic Sinus Surgery (ESS). Investigators want to understand how adding a medication called dupilumab to their usual treatment affects inflammation in their upper and lower airways over 24 weeks.

Dupilumab works by blocking certain signals in the immune system that contribute to inflammation in both the sinuses and the lungs. By studying how this medication changes the immune profiles of both airway systems, investigators hope to learn more about the underlying causes of airway inflammation in these conditions.

This research is important because it may help understand if treating inflammation in one part of the airway (like the lungs) has a similar effect on inflammation in another part (like the sinuses). This could lead to better treatments for people with CRSwNP and asthma, targeting the root causes of their symptoms more effectively.

DETAILED DESCRIPTION:
In adult patients with CRSwNP with concomitant moderate-severe asthma undergoing Endoscopic Sinus Surgery (ESS), what is the change in the inflammatory cascade in the upper and lower airways from patients treated with 300 mg of dupilumab twice daily for 24 weeks as an add-on treatment to the standard of care (intranasal corticosteroids, INCS+ backgroung asthma medication) compare to the placebo + standard of care treatment only.

The investigators hypothesize that the study of the immune profile in patients with CRSwNP and asthma would give a better understanding of the mechanism involved in the airway inflammatory response. Determining the molecular profiles of the upper and lower airways after dupilumab treatment has not been studied yet.

Dupilumab has demonstrated effectiveness in treating both Chronic Rhinosinusitis with Nasal Polyps (CRSwNP) and asthma, conditions characterized by Type 2 inflammation, by inhibiting the IL-4 and IL-13 signalling pathways. However, it remains unclear how immunological changes occur in paired tissues of the upper (sinus) and lower (lung) airways in patients treated with biologics compared to those receiving standard therapies. Additionally, it is not well understood whether improvements in one airway system (e.g., the lungs) are mirrored in the other (e.g., the sinuses), which could result in differing clinical responses. This study aims to address these gaps by examining the comparative effects of Dupilumab versus standard treatments on both airway systems, to determine if therapeutic effects are consistently observed across both systems and to understand the potential implications for clinical responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 19.
* Patients undergoing Endoscopic Sinus Surgery (ESS)
* Patients with CRSwNP with moderate-severe asthma according to 2020 EPOS criteria:

  1. Asthma confirmed with spirometry and assessment on the previous history of asthma (a methacholine challenge test and atopy testing to document the positive or negative history of asthma will be performed if there is no clinical record). Asthma severity based on GINA guidelines.
  2. Presence of nasal polyps. This can be based on the formal exam at Baseline Visit or historical assessment.

Exclusion Criteria:

* Patients with current or past sinonasal or bronchial tumours
* Subjects who have been treated with oral antibiotics in the past month prior to surgery
* Subjects with known immunodeficiency
* Subjects with known autoimmune disease
* Subjects with other sinonasal diseases other than CRSwNP (e.g., cystic fibrosis, eosinophilic granulomatosis with polyangiitis, allergic fungal rhinosinusitis, invasive fungal sinusitis, fungal ball, dyskinetic cilia syndrome)
* Prior lung transplants
* Subjects with hypersensitivity; with allergy/intolerance to a monoclonal antibody or biologic
* Prior use of dupilumab or other biologic medications (omalizumab. mepolizumab, reslizumab,etc) 6 months before enrollment.
* Any condition that, in the opinion of the investigator, may interfere with the patient's ability to participate in the study per protocol.
* Participation in an ongoing interventional or observational study using a biologic treatment.
* Female participants who are pregnant or breastfeeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Cytokine levels such as GM-CSF, IFNg, TNFa, VEGF-A, Identification of Key Interleukins and chemokynes (10/CXCL10, MIP-1a/CCL3, RANTES/CCL5), compared with placebo in CRSwNP and asthma patients from baseline to week 24 | From baseline to 24 weeks.
  Change in GM-CSF, IFNg, IL-1b, IL-2, IL-4, IL-5, IL-6, IL-8, IL-10, IL-12 (p40), IL-13, IL-17A, IP-10/CXCL10, MIP-1a/CCL3, RANTES/CCL5, TNFa, VEGF-A compared with placebo in CRSwNP and asthma patients from baseline to week 24

SECONDARY OUTCOMES:
Changes in SNOT-22, ACQ-5 and Sniffin Stick Test | 24 weeks
  Relation of changes in the inflammatory profiles with changes in symptom control (SNOT-22, ACQ-5,Sniffin Stick test) compared with placebo at baseline and 24 weeks.
Relation of changes in inflammatory profile with changes in endoscopic scores (MLK) | 24 weeks
  Correlate the changes in the inflammatory profiles with changes in endoscopy scores (MLK scores) compared with placebo at baseline and 24 weeks.
Relation of inflammatory profile and (FeNO and nasal FeNO) | 24 weeks
  Correlate the changes in the inflammatory profiles with changes in the pulmonary function measured by spirometry FEV1 values and standard and nasal fractional exhaled nitric oxide (FeNO and nasal FeNO) compared with placebo at baseline and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Thamboo, Principal Investigator — St Paul's Sonis Centre Director

IPD SHARING:
Plan to Share IPD: No